CLINICAL TRIAL: NCT05588453
Title: A Phase I/II Study of Ex-Vivo Expanded Allogeneic Universal Donor (UD) TGFbi NK Cell Infusions in Combination With Temozolomide as a Lymphodepleting Agent in Patients With Melanoma Metastatic to the Brain
Brief Title: Natural Killer Cell Therapy (UD TGFbetai NK Cells) and Temozolomide for the Treatment of Stage IV Melanoma Metastatic to the Brain
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kari Kendra (Other)
Responsible Party: Sponsor-Investigator, Kari Kendra, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21101; NCI-2021-14033 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-09-05; First posted 2022-10-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (UD TGFbetai NK cells, temozolomide) (Experimental): Patients receive UD TGFbetai NK cells IV over 30 minutes on day 1 and temozolomide PO daily on days 1-5. Treatment with UD TGFbetai NK cells repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Cycles of temozolomide repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Natural Killer Cell Therapy; Drug: Temozolomide

INTERVENTIONS:
Biological: Natural Killer Cell Therapy — Given UD TGFbi NK cell IV
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of universal donor UD TGFbetai natural killer (NK) cells, and whether UD TGFbetai NK cells with temozolomide works to shrink tumors in patients with stage IV melanoma that has spread to the brain (metastatic to the brain). NK cells are immune cells that contribute to anti-tumor immunity by recognizing and destroying transformed or stressed cells. Temozolomide is in a class of medications called alkylating agents. It works by slowing or stopping the growth of cancer cells in the body. Giving UD TGFbetai NK cell and temozolomide may work better in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm the safety and tolerability of UD TGFbetai NK cells in combination with temozolomide as a lymphodepleting agent in patients with melanoma metastatic to the brain and to determine the recommended phase 2 dose (RP2D). (Phase 1) II. To determine the intracranial response rate. (Phase 2)

SECONDARY OBJECTIVES:

I. To define the toxicities of UD TGFbetai NK cells when delivered with temozolomide as a lymphodepleting agent. (Phase 1) II. To define the pharmacokinetics (pK) associated with UD TGFbetai NK cells when used in combination with temozolomide as a lymphodepleting agent in patients with metastatic melanoma. (Phase 1) III. To determine the extracranial response rate. (Phase 2) IV. To determine progression free survival (PFS) (intracranial, extracranial, overall). (Phase 2) V. To assess overall survival (OS). (Phase 2) VI. To continue to assess the safety of temozolomide in combination with UD TGFbetai NK cells in a patient with melanoma metastatic to the brain. (Phase 2)

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. To assess the phenotype and function of the UD TGFbetai NK cells and correlate with clinical outcomes.

II. To assess in vivo persistence of UD TGFbetai NK cells after adoptive transfer and correlate with clinical outcomes.

III. To assess immune status, inflammatory cytokine levels, and anti-melanoma cell activity.

OUTLINE: This is a phase I, dose-escalation study of UD TGFbetai NK cells followed by a phase II study.

Patients receive UD TGFbetai NK cells intravenously (IV) over 30 minutes on day 1 and temozolomide orally (PO) daily on days 1-5. Treatment with UD TGFbetai NK cells repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Cycles of temozolomide repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma with stage IV disease
* Radiologically confirmed brain metastasis (n >= 1) with at least one measurable central nervous system (CNS) lesion >= 10 mm on T1-weighted gadolinium enhanced magnetic resonance imaging (MRI) and unequivocal evidence of progression
* No indication for stereotactic radiotherapy
* At least 4 weeks from any anticancer treatment (cytotoxic chemotherapy, signal transduction inhibitors, immunotherapy or radiation)
* Absolute neutrophil count (ANC) 1 x 10^9/L
* Platelets > 100,000/L
* Hemoglobin (Hgb) >= 10 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Albumin >= 2.5 g/dL
* Serum bilirubin < 1.5 x ULN unless due to Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN if documented liver metastases or < 3 X ULN without liver metastasis
* > 18 years old (y/o)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Females of reproductive age must agree to the use of an effective contraceptive method while on treatment, beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product for women. Males able to father a child must practice adequate methods of contraception or completely abstain from intercourse from the first dose of investigational treatment until one week after the final dose of investigational treatment
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of enrollment and/or urine pregnancy test 48 hours prior to the administration of the first study treatment
* Patient information and written informed consent form signed

Exclusion Criteria:

* Planned or concurrent systemic treatment or radiation therapy
* If requiring corticosteroids for cerebral edema, patients must be on a stable dose. Lowest dose of steroids needed to control CNS edema is recommended. Doses above 4 mg daily need to be cleared by principal investigator (PI) of the study
* Known contra-indication to MRI
* Patients with non-melanoma malignancies are excluded unless a complete remission has been achieved at least 3 years prior to study entry and no additional therapy is required or anticipated during the study period (exceptions include: non-melanoma skin cancers, in situ bladder cancer, in situ gastric cancer, in situ colon cancers, in situ cervical cancers/dysplasia, or in situ breast carcinoma)
* Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as:

  * Active infection
  * Current active hepatic or renal disease
  * Pregnant women, women who are likely to become pregnant or are breastfeeding
  * Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological, or geographical conditions potentially hampering ability to consent, compliance with the study protocol, and follow-up schedule; those conditions should be discussed with the patient before remigration in the trial
  * Patients who received any other investigational drugs within the 30 days prior to screening visit
  * Leptomeningeal metastases diagnosed by MRI
  * Inclusion in another therapeutic protocol within 30 days
  * If steroids are necessary to control symptoms related to CNS metastases, patients should be on the lowest dose of steroids necessary to control symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities (Phase I) | Up to 28 days
  Toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 4.03. The CTCAE provides descriptive terminology and a grading scale for each adverse event listed. All toxicities will be summarized as the percentage of patients experiencing each type and grade of event according to dose level.
Incidence of adverse events (AEs) (Phase I) | Up to 5 years
  Assessed using CTCAE version (V)4.0. All toxicities will be summarized as the percentage of patients experiencing each type and grade of event according to dose level. Patients who receive at least one dose of treatment will be included in the analysis. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Proportion of subjects who achieve an intracranial complete response or partial response (Phase II) | Up to 5 years
  Assessed using modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.

SECONDARY OUTCOMES:
Incidence of adverse events of universal donor (UD) TGFbetai natural killer (NK) cells when delivered with temozolomide as a lymphodepleting agent (Phase I) | Up to 5 years
  Assessed using CTCAE V5.0. All toxicities will be summarized as the percentage of patients experiencing each type and grade of event according to dose level. Patients who receive at least one dose of treatment will be included in the analysis. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Extracranial response rate (Phase II) | Up to 5 years
  Assessed using RECIST criteria. Will be calculated as the proportion of patients who achieve a response to therapy divided by the total number of evaluable patients. An evaluable patient is defined as an eligible patient who has received at least one dose of therapy. All evaluable patients will be included in calculating the response rate for the study along with corresponding 95% binomial CIs (assuming that the number of patients who respond is binomially distributed).
Progression free survival (PFS) (intracranial, extracranial, overall) (Phase II) | From initiation of therapy to the time of Response Evaluation Criteria in Solid Tumors (RECIST) progression or death, assessed up to 5 years
  Survival will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% confidence interval (CI), assuming sufficient events have occurred.
Overall Survival (OS) (Phase II) | From initiation of therapy to death, assessed up to 5 years
  Survival will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Percentage of patients with adverse events of the combination temozolomide and UD TGFbetai NK cells (Phase II) | Up to 5 years
  The percentage of patients with adverse events as assessed by CTCAE V 5.0 criteria. Frequency and severity of AEs will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns
Pharmacokinetics (PK) parameters associated with UD TGFbetai NK cells (Phase I) | Within 1 hour prior to UD TGFbetai NK infusions and within 30 minutes post infusion on cycle 1, day 15 (C1D15), C1D17, and C1D19] and prior to cycle 2 day 1 and cycle 3 day 1. (Each cycle is 28 days)
  The samples will be analyzed using the Devyser Chimerism assay to identify the UD TGFbeta iNK cells. We will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations [GEE]) to assess the PK described above in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.

OTHER OUTCOMES:
Phenotype and function of the UD TGFbetai NK cells | Up to 5 years
  Will be correlated with clinical outcomes. Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean +/- standard error of the mean (SEM), range, and median at each time point. Associations with clinical outcomes will be evaluated using two-sample t test or Fisher exact test.
Persistence of UD TGFbetai NK cells | Up to 5 years
  Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean +/- SEM, range, and median at each time point. Associations with clinical outcomes will be evaluated using two-sample t test or Fisher exact test.
Distribution of UD TGFbetai NK cells in the cerebrospinal fluid (CSF) | Up to 5 years
  Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean +/- SEM, range, and median at each time point. Associations with clinical outcomes will be evaluated using two-sample t test or Fisher exact test.
Immune activation post infusion | Up to 5 years
  Graphical analyses will be largely used to assess potential patterns and relationships. All continuous measurements will be summarized using mean +/- SEM, range, and median at each time point. Associations with clinical outcomes will be evaluated using two-sample t test or Fisher exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Kari L Kendra, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu